CLINICAL TRIAL: NCT02919839
Title: Measuring and Predicting Glycemic Response to Food in Patients With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Orit Hamiel (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor-Investigator, Dr. Orit Hamiel, Director of the Pediatric Endocrinology and Diabetes Unit, Sheba medical center, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: 2.0
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Personalized Medicine in Type 1 Diabetes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood glucose, microbiome
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non-Interventional

SUMMARY:
Personalized medicine methods in the management of type 1 diabetes

DETAILED DESCRIPTION:
This proposal joins together clinical practitioners, biologists, and computer scientists to set up the infrastructure for research that will facilitate, for the first time, the use of big-data, machine-learning approaches in the application of personalized medicine methods in the management of type 1 diabetes mellitus. We will model the clinical, microbial, and nutritional factors underlying the variability in glycemic response to food in this population; develop algorithms for prediction of this response and for the accurate administration of insulin, assisting the clinical management of the disease and discover intervention targets in the gut microbiome aimed at improving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

over one year of diagnostic with T1DM.

Exclusion Criteria:

Drug related diabetes. genetical diabetes.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
blood glucose | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orit Hamiel, Prof, Principal Investigator — Sheba Medical Center; Eran Segal, Prof., Principal Investigator — Weizmann Institute of Science

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shilo S, Godneva A, Rachmiel M, Korem T, Bussi Y, Kolobkov D, Karady T, Bar N, Wolf BC, Glantz-Gashai Y, Cohen M, Zuckerman-Levin N, Shehadeh N, Gruber N, Levran N, Koren S, Weinberger A, Pinhas-Hamiel O, Segal E. The Gut Microbiome of Adults With Type 1 Diabetes and Its Association With the Host Glycemic Control. Diabetes Care. 2022 Mar 1;45(3):555-563. doi: 10.2337/dc21-1656. PMID 35045174
- [Derived] Shilo S, Godneva A, Rachmiel M, Korem T, Kolobkov D, Karady T, Bar N, Wolf BC, Glantz-Gashai Y, Cohen M, Zuckerman Levin N, Shehadeh N, Gruber N, Levran N, Koren S, Weinberger A, Pinhas-Hamiel O, Segal E. Prediction of Personal Glycemic Responses to Food for Individuals With Type 1 Diabetes Through Integration of Clinical and Microbial Data. Diabetes Care. 2022 Mar 1;45(3):502-511. doi: 10.2337/dc21-1048. PMID 34711639